CLINICAL TRIAL: NCT02713945
Title: Treatment With HMG-COA Reductase Inhibitor (Simvastatin) of Growth and Bone Abnormalities in Children With Noonan Syndrome: A Phase III Randomised, Double Blind, Placebo-controlled Therapeutic Trial
Brief Title: Treatment With HMG-COA Reductase Inhibitor of Growth and Bone Abnormalities in Children With Noonan Syndrome
Acronym: RASTAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/15/7826
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Noonan Syndrome
Keywords: Simvastatin; Ras; MAPK
MeSH Terms: conditions — Noonan Syndrome | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin administrated orally at 10 mg once a day in the morning during the first month Simvastatin administrated orally at 20 mg once a day in the morning during the second month During months 3 to 12, the dose will be fixed at 20 mg per day for children aged 12 years and younger and 40 mg for adolescent older than 12 years.
  Interventions: Drug: Simvastatin
- Control (Placebo Comparator): Placebo administrated orally once daily in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Experimental drug administrated orally
  Arms: Simvastatin
Drug: Placebo — Treatment for the control group
  Arms: Control

SUMMARY:
This study evaluate the efficacy of 3-hydroxy-3-methylglutaryl coenzyme A (HMG-COA) reductase inhibitors, also known as "statins" in the treatment of growth and skeletal abnormalities in children with Noonan syndrome. Half of patients will receive simvastatin while the other half will receive a placebo.

DETAILED DESCRIPTION:
Noonan syndrome (NS) is a relatively frequent autosomal dominant disorder characterised by facial dysmorphic features, heart defects, developmental delay, and short stature. This syndrome is mostly caused by gain-of-function mutations in the PTPN11 gene, encoding tyrosine phosphatase. The best-defined consequence of NS-causing mutants is an enhancement of Ras/MAPK activation that is responsible for the different NS features. Mutations in several genes encoding other components of the Ras/Mitogen Activated Protein Kinase (MAPK) pathway, resulting in hyperactivation, are also found in syndromes close to NS.

Short stature caused by growth hormone insensitivity and skeletal abnormalities are major concerns in NS. To date there is no effective specific therapy for affected patients. Given the role of Ras/Mitogen Activated Protein Kinase (MAPK) activation in NS pathophysiology, therapeutic strategies aiming to reduce this activation seem to be very promising.

Recently, 3-hydroxy-3-methylglutaryl coenzyme A (HMG-COA) reductase inhibitors, also known as "statins" have been suggested as a potential therapy by decreasing Ras activity.

The efficacy of statins for treating cognitive deficits have been reported in mouse models of NS. Statins (simvastatin) have been assessed in mouse models and clinical studies for the treatment of cognitive deficits in children with discordant results but good tolerance. Recently, it has been demonstrated that statins may also correct bone growth abnormality in a mouse model for achondroplasia.

As growth is usually normal at birth in NS patients and thereafter progressively worsens throughout childhood, the investigators expect that precocious modulation of Ras/MAPK activation by statins may attenuate growth retardation. To achieve this goal, the present study is the first prospective randomised placebo-controlled therapeutic trial using statins in children with NS.

Marketing authorisation for statins is already accepted for the treatment of children with familial hypercholesterolemia and worldwide marketing authorisation of statins.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Noonan syndrome
* Female child between 6 to 15 years, without menses, with bone age < 13 years
* Male child between 6 to 16 years, with bone age < 14 years
* Decreased growth velocity (< -1 SDS) and/or short stature (height < -2 SDS or -1,5 SDS under target height)
* Informed consent obtained from child and parents

Exclusion Criteria:

* Contraindication to simvastatin treatment :
* Progressive liver disease, increased serum levels of alanine aminotransferase (ALT) (> 1,5 uper limit of normal (ULN)), aspartate aminotransferase (> 1,5 ULN)
* Known hypersensitivity to simvastatin
* Pregnancy
* Treatment with CYP3A4 inhibitors (erythromycin, clarithromycin, ketoconazole, or itraconazole)
* Growth promoting therapies such as recombinant human Growth Hormone (GH) or IGF-1 treatment

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Effect of a 12-month simvastatin treatment on growth in NS children as assessed by change in Insulin-like Growth Factor-1 (IGF-1) levels converted to age and sex specific z-scores | Baseline, month 1, month 3, month 6, month 9 and month 12

SECONDARY OUTCOMES:
Effect of a 12-month simvastatin treatment on growth velocity as assessed by Height measurement. | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on body mass index as assessed by height and weight measurement. | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on waist circumference as assessed by clinical examination | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on hormonal growth parameters as assessed by serum IGFBP-3 levels | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on growth plates as assessed by serum C-type natriuretic peptide (CNP) levels | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on growth plates as assessed by serum amino-terminal propeptide of CNP (NTproCNP) levels | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on bone formation as assessed by serum bone alkaline phosphatase (BAP) levels | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on bone resorption as assessed by serum carboxy-terminal collagen crosslinks (CTX) levels | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on cardiac function as assessed by echocardiography | Baseline and month 12
Effect of a 12-month simvastatin treatment on cognitive deficits as assessed by parent-rated child behaviour checklist (CBCL) | Baseline and month 12
Effect of a 12-month simvastatin treatment on behavioural deficits as assessed by parent-rated child behaviour checklist (CBCL) | Baseline and month 12
Effect of a 12-month simvastatin treatment on metabolism of lipids as assessed by lipids levels. | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on metabolism of lipids as assessed by leptin levels. | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on metabolism of lipids as assessed by adipokines levels. | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on fat body mass as assessed by Dual-energy X-ray Absorptiometry (DXA). | Baseline and month 12
Effect of a 12-month simvastatin treatment on insulin sensitivity indices as assessed by Homeostasis Model Assessment of Insulin Resistance (HOMA-IR). | Baseline, month 1, month 3, month 6, month 9 and month 12
Effect of a 12-month simvastatin treatment on insulin sensitivity indices as assessed by Quantitative Insulin-Sensitivity Check Index (QUICKI) | Baseline, month 1, month 3, month 6, month 9 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Edouard, MD, PHD, Principal Investigator — Children's Hospital, Toulouse University Hospital
Locations (12):
- France (12):
  - CHU Angers Unité d'endocrinologie pédiatrique, Angers
  - CHU Bordeaux Unité de Génétique pédiatrique, Bordeaux
  - Chu Dijon, Dijon
  - CHRU Lille Unité d'endocrinologie pédiatrique, Lille
  - CHU Lyon Unité d'endocrinologie pédiatrique, Lyon
  - CHU Marseille La Timone Unité d'Endocrinologie pédiatrique, Marseille
  - Chu Montpellier, Montpellier
  - CHU Nancy Unité de Génétique pédiatrique, Nancy
  - Hôpital Robert Debré Unité de Génétique pédiatrique, Paris
  - Hôpital Trousseau Unité d'endocrinologie pédiatrique, Paris
  - CHU Rennes Unité de Génétique pédiatrique, Rennes
  - CHU Toulouse Hôpital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No